CLINICAL TRIAL: NCT03955822
Title: Essure Permanent Birth Control, Effectiveness and Safety: A French Survey
Acronym: prevessure
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018-843-0025
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Contraception
Keywords: effectiveness; security; adverse effects; permanent birth control

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Phone survey — Phone Survey in order to evaluate adverse effect of the permanently implanted birth control device for women (Essure) will be proposed to wmen Treated between 2002 and 2017 with Essure.

SUMMARY:
Since 2002, in CHU Amiens, Essure implants started to be used for women in need of voluntary sterilization in accordance with French national recommendations. Recently patient committees emerged to alert health agency and governments about various symptoms possibly link to the Essure implants. New studies have been launched in order to determinate if Essure implants were involved with the symptoms described. According to the scientific literature no solid link between Essure and the symptomatology was highlighted. French National College of Gynecologists and Obstetricians send a letter of information for patient and gynecologists. French National agency of medicament suspended Essure authorization in august 2017 for 3 months. Bayer industry decided to withdraw from the market the Essure implants in autumn 2017. Currently Essure procedures have been stopped to be used in CHU Amiens since august 2017. But, in CHU Amiens, health institutions still have to manage patients with Essure implants and potential adverse effects.

The purpose of this study is to determine if the patients treated between 2002 and 2017 with Essure implant present complications, had a proper follow up after the Essure implantation, and that the Essure implantation respected the medical guidelines in order to offer the best medical care with these new informations.

Medical data from patients who received Essure procedure will be collected with medical file and a survey about adverse effects will be submitted to patients by phone if they agree to take part of the study after loyal information.

ELIGIBILITY:
Inclusion Criteria:

* women more than 18 years old
* patients who benefit of Essure permanent birth control in CHU Amiens between 2002 and 2017
* signed informed consent form

Exclusion Criteria:

* women Under 18 years old
* refusal to participate
* patient Under administrative supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who underwent volontary sterilization with the Essure implant
Study Population: Women who underwent volontary sterilization with the Essure permanent birth control in CHU Amiens between 2002 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Number of side effects of Essure system for the patient | patients who benefited of Essure implant between 2002 and 2017
  this outcome is evaluated with data of medical files and with a phone survey submitted to the patient who had the essure procedure in CHU Amiens.

SECONDARY OUTCOMES:
Number of patients who underwent Essure implant withdrawal | between 2002 and day of patient inclusion
  this outcome is evaluated with data of medical files and with a phone survey

CONTACTS AND LOCATIONS:
Overall Officials: fabrice sergent, Pr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No